CLINICAL TRIAL: NCT01390077
Title: Nitisinone (NTBC) In Different Age Groups Of Patients With Alkaptonuria
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WLN02
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Alkaptonuria
Keywords: homogentisic acid
MeSH Terms: conditions — Alkaptonuria | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitisinone (Experimental): all subjects will receive open-label nitisinone
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — Taken orally. Supplied as a 2mg tablet. The starting dose is 2 mg once daily.
  Other Names: Orfadin®,; NTBC

SUMMARY:
Nitisinone is a potent inhibitor of the enzyme that catalyzes the formation of homogentisic acid, and should be an even more logical treatment for alkaptonuria than for tyrosinemia, for which it has been approved by the FDA.The objective of this research is to explore reported age related differences in toxicity of nitisinone and its pharmacokinetic underpinnings and to develop an optimal therapeutic requirement for a targeted population of presymptomatic patients. The additional effect of mixtures of amino acids excluding tyrosine will be explored to take advantage of protein synthesis to avoid elevations of tyrosine that would otherwise limit the optimal dosage of nitisinone. The study is designed to treat patients and find the optimal dosage of nitisinone to obtain maximal reduction in levels of homogentisic acid and maintain safe levels of tyrosine.

The long term objective in the target population of pre-symptomatic patients is the prevention of the characteristic effects on joint cartilage and tendons.

DETAILED DESCRIPTION:
Study procedures are designed to:

1. Develop a method for nitisinone measurement via tandem mass spectrometry (MS/MS).
2. Determine whether differences between adult and children could be erased by employing a dosage regimen based on m2 of body surface area as opposed to per kg of body weight, as we have found in a recent study of dichloroacetate
3. Determine optimal dosage for reduction of urinary levels of homogentisic acid and minimal elevation of plasma levels of tyrosine in the target population of pre-symptomatic patients.
4. Determine optimal doses of Tyrex to prevent hypertyrosinemia and allow maximal reduction in homogentisic acid.

Baseline studies will include ophthalmologic examinations, echocardiogram, X-rays of all joints, MRI of selected joints when financially plausible; history and physical examinations with emphasis on joints and tendons. Ideally MRI will be repeated at 12 month intervals thereafter. Ophthalmologic exam, x-rays of the kidneys and prostate, and echocardiogram will be repeated approximately every 12 months, depending on the age of the subject and the nitisinone dose. Patients will be seen every 3 months for the first year, then at 6 month intervals to month 36. The timing of the visits may be altered in response to modifications of nitisinone and/or Tyrex doses.

Complete or near complete elimination of homogentisic acid excretion will be sought. Optimal NTBC dosage would be judged to yield plasma concentration of tyrosine less than 1000 mmol/L with the concomitant use of tyrosine free amino acid supplement. Dosage will be escalated or reduced dependent on evidence of accumulation of nitisinone and urinary levels of HGA. The maximum initial dose of nitisinone for adult and adolescent patients will be 0.2/mg/kg/day, younger patients may require a larger dose; the standard dose in hypertyrosinemia is 1mg/kg/day, which will be tentatively used as the maximum dose for all populations.

Patients will be asked to collect first morning or 12 hour urine collections for homogentisic acid and p-hydroxyphenyllactic acids and to monitor levels of tyrosine. Accumulation will be tested for by repeated studies after 3 months of treatment. Trough levels for nitisinone will be collected prior to and 5-7 days after dose increases and/or at months 6, 12, 18, 24 and every 12 months.

The SF-36 Health Status Survey, a two page quality of life questionnaire which asks about ADLs and emotional/social impacts of disease, will be completed by the patient or patient's parent at baseline and every six months.

At any point during the study if the plasma tyrosine level is greater than 900umol/L the amount of Tyrex or dietary protein intake may be modified, or the nitisinone dose may be decreased. Protein Saver blood spot cards, which can be done in the patient's home and mailed to our lab, will be given to the patients with instructions on blood collection to check the tyrosine level after 5-7 days of the drug/dietary modifications. These steps-the dietary modification with diet records if needed, addition or adjustment of Tyrex, adjustment of the nitisinone dose, and repeat tyrosine analysis-will be repeated as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of alkaptonuria with documented increased excretion of homogentisic acid
2. Willing and able to provide written, signed informed consent, or age appropriate written assent and written informed consent by a legally authorized representative after the study has been explained, prior to any research-related procedures.
3. Willing and able to be seen in the UCSD Clinical Center for Research or a satellite site for the study visits
4. Possession of insurance coverage for standard of care procedures, clearly stated in the consent forms

Exclusion Criteria:

1. Baseline tyrosine level above 250 mmol/mL
2. Baseline serum creatinine, creatine kinase, or transaminases 2x upper limit of normal
3. Baseline anemia or thrombocytopenia
4. Current participation in another investigational medication trial.
5. Pregnant or lactating women
6. Current keratopathy, contact use or uncontrolled glaucoma
7. History myocardial infarction or arrhythmia
8. History of pulmonary insufficiency
9. Psychiatric illness that may interfere with compliance or communication
10. Current malignancy or hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Nyhan, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Suwannarat P, O'Brien K, Perry MB, Sebring N, Bernardini I, Kaiser-Kupfer MI, Rubin BI, Tsilou E, Gerber LH, Gahl WA. Use of nitisinone in patients with alkaptonuria. Metabolism. 2005 Jun;54(6):719-28. doi: 10.1016/j.metabol.2004.12.017. PMID 15931605
- [Background] Introne WJ, Perry MB, Troendle J, Tsilou E, Kayser MA, Suwannarat P, O'Brien KE, Bryant J, Sachdev V, Reynolds JC, Moylan E, Bernardini I, Gahl WA. A 3-year randomized therapeutic trial of nitisinone in alkaptonuria. Mol Genet Metab. 2011 Aug;103(4):307-14. doi: 10.1016/j.ymgme.2011.04.016. Epub 2011 May 6. PMID 21620748
- [Background] Phornphutkul C, Introne WJ, Perry MB, Bernardini I, Murphey MD, Fitzpatrick DL, Anderson PD, Huizing M, Anikster Y, Gerber LH, Gahl WA. Natural history of alkaptonuria. N Engl J Med. 2002 Dec 26;347(26):2111-21. doi: 10.1056/NEJMoa021736. PMID 12501223
- [Background] Gertsman I, Gangoiti JA, Nyhan WL, Barshop BA. Perturbations of tyrosine metabolism promote the indolepyruvate pathway via tryptophan in host and microbiome. Mol Genet Metab. 2015 Mar;114(3):431-7. doi: 10.1016/j.ymgme.2015.01.005. Epub 2015 Jan 29. PMID 25680927
- [Result] Gertsman I, Barshop BA, Panyard-Davis J, Gangoiti JA, Nyhan WL. Metabolic Effects of Increasing Doses of Nitisinone in the Treatment of Alkaptonuria. JIMD Rep. 2015;24:13-20. doi: 10.1007/8904_2014_403. Epub 2015 Feb 10. PMID 25665838

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitisinone: All subjects received open-label nitisinone, taken orally, supplied as a 2mg tablet. The starting dose was 2 mg once daily, and increased to 4, 6, or 8 mg, case-by-case.
Period: Overall Study
Arm/Group | Nitisinone
Started | 8
Treatment | 7
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 8 patients consented; only 7 continued to treatment.
Arm/Group | Nitisinone
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 47 [31 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Homogentisic Acid Excretion
Description: Urine homogentisic acid (umol/mmol creatinine)
Time Frame: 3-6 months
Measure: Mean (Standard Deviation); unit: uM
Groups:
- HGA, Baseline: Urine homogentisic acid (umol/mmol Cr), while taking no nitisinone
- HGA, 2 mg/d Nitisinone: Urine homogentisic acid (umol/mmol Cr), while on nitisinone, 2 mg/d
- HGA, 4 mg Nitisinone: Urine homogentisic acid (umol/mmol Cr), while on 4 mg/d nitisinone
Arm/Group | HGA, Baseline | HGA, 2 mg/d Nitisinone | HGA, 4 mg Nitisinone
Number analyzed (Participants) | 7 | 7 | 6
uM | 1425.9 (678.3) | 113.1 (70.9) | 34.0 (12.9)

2. Secondary Outcome: Tyrosine Levels
Description: Plasma tyrosine (uM)
Time Frame: 3-6 months
Measure: Mean (Standard Deviation); unit: uM
Groups:
- Tyrosine, Baseline: Plasma tyrosine (uM), while taking no nitisinone
- Tyrosine, 2 mg/d Nitisinone: Plasma tyrosine (uM), while on nitisinone, 2 mg/d
- Tyrosine, 4 mg Nitisinone: Plasma tyrosine (uM), while on 4 mg/d nitisinone
Arm/Group | Tyrosine, Baseline | Tyrosine, 2 mg/d Nitisinone | Tyrosine, 4 mg Nitisinone
Number analyzed (Participants) | 7 | 7 | 6
uM | 53.1 (14.8) | 668.7 (114.7) | 703.7 (120.8)

ADVERSE EVENTS:
Time Frame: Patients were monitored up to 3.5 years. Patients 1-3 were monitored over the course of 3-3.5 years, while patients 4-7 were monitored between 0.5 and 1 year
Groups:
- Nitisinone: All subjects who participated in treatment received open-label nitisinone, taken orally, supplied as a 2mg tablet.
  The starting dose was 2 mg once daily, and increased to 4, 6, and 8 mg/d, case-by-case.
Arm/Group | Nitisinone
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitisinone (N=7)
Ocular irritation (Eye disorders) | 2 — Eye discomfort and blurry vistion
Abdominal discomfort (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes